CLINICAL TRIAL: NCT00582569
Title: Breast MRI Spectroscopy, Department of Defense (DOD)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 05-101
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Breast Lesion
Keywords: Breast lesion; Spectroscopy; MRI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this new imaging method is to provide physicians with additional information not available with standard imaging methods. This includes information about the make up of different breast diseases. Using spectroscopy data, it may be possible to tell the difference between benign conditions of the breast from malignant tumors and provide more accurate information than can be obtained with regular MRI. Along with the MRI a new method of evaluating the images or pictures will be used. This new method is called spectroscopy and is used routinely on other parts of the body such as the prostate and brain. Pictures produced with this sequence look different than the regular MRI pictures. Performing spectroscopy on a 1.5T magnet adds another imaging sequence (another scan) to the routine MRI protocol, thus increasing exam time (extra 10-15 minutes). This study will enroll patients who are scheduled for a Magnetic Resonance Imaging (MRI) examination ordered by their primary physician.

DETAILED DESCRIPTION:
Our aim is to perform MR Spectroscopy (MRS) on 150 patients at the end of their clinically indicated routine breast MRI guided biopsy and breast MRI guided needle localization examination using a software package from General Electric Medical Systems (Milwaukee,WI). This will add time to the routine examination but will not involve additional injections of contrast. We will analyze the spectroscopic data to determine if benign lesions can be reliably differentiated from malignant ones. The MR Spectroscopy (MRS) will be administered at Memorial Sloan Kettering Cancer Center, 1275 York Ave, NY,NY 10021.

ELIGIBILITY:
Inclusion Criteria:

* Patient needs to be ≥ or = to 18 years of age
* scheduled for diagnostic breast MRI examination or interventional procedure for a suspected or known breast lesion ≥ or = to 1 centimeter

Exclusion Criteria:

* Patients who would be normally excluded from undergoing an MRI examination include:
* Patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field
* Patients who are pregnant are excluded from participation of this study
* Patients who are unable to comply or complete the MRI exam due to claustrophobia or high levels of anxiety.
* Patients undergoing chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Include women with lesions, > or = to 1 centimeter that will undergo a diagnostic MRI exam, an MRI guided biopsy, or an MRI guided needle localization, such as women with breast cancer or women with clinical and/or mammographic findings suspicious for breast masses. However, any known breast lesion, benign or malignant, will be appropriate for evaluation with MR spectroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2006-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
to determine if spectroscopy of the breast can be performed and can be functional in a clinical environment for breast lesions _> 1centimeter | conclusion of study
To see if MRS can differentiate ben vs mal breast tissue with adequate specificity & sensitivity to be useful in clinical management. | conclusion of study

SECONDARY OUTCOMES:
if the data obtained can differentiate among various histologic subtypes of invasive and non-invasive breast cancers, and can be reliably analyzed and be useful to the final interpretation of the breast MRI examination. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Brennan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center website — http://www.mskcc.org